CLINICAL TRIAL: NCT02827370
Title: CAREFOR Study: Precision Nutrition Caloric Restriction for Oncology Research: Precision Medicine Driving Precision Nutrition During Neoadjuvant Chemotherapy for Breast Cancer
Brief Title: CAREFOR: Precision Medicine Driving Precision Nutrition for the Treatment of NeoAdjuvant Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16D.067; JT 8562 (Other: JeffTrial Number)
Record Dates: First submitted 2016-06-13; First posted 2016-07-11 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Precision Nutrition (dietary intervention) (Experimental): During chemotherapy, patients will receive dietary counseling based on the molecular pathways driving their specific breast cancers found through genetic testing. Nutritional recommendations will seek to down-regulate the dominant molecular drivers of an individual's breast cancer while they are receiving standard chemotherapy as outlined by their treating medical oncologist.
  Interventions: Behavioral: Behavioral Dietary Intervention

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Receive dietary counseling

SUMMARY:
The purpose of the study is to determine if a targeted dietary change can enhance the effect of neo-adjuvant chemotherapy

DETAILED DESCRIPTION:
Primary objective:

I To determine if dietary alternations designed to downregulate the dominate molecular drivers of an individuals' breast cancer will enhance the effect of neoadjuvant chemotherapy and allow for an increase in the pathologic complete response rate.

Secondary objectives

I) Investigator measurable changes to molecular and patient characteristics from precision nutrition to determine a metric for evaluation this treatment in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven invasive breast cancer
* Planned neoadjuvant chemotherapy determined by the judgment of the medical oncologist
* The patient must be female
* Age ≥ 18
* Non-metastatic and non-inflammatory breast cancer
* History/physical examination, including breast exam and documentation of weight and Karnofsky Performance Status of 80-100% for at least 60 days prior to study entry.
* Women of childbearing potential must be non-pregnant and non-lactating and willing to use medically acceptable form of contraception during chemotherapy
* Patient must capable of and provide study specific informed consent prior to study entry
* BMI ≥21
* Weight ≥120lbs
* No prior history of non-breast malignancies in the past 1 year unless it was a non- melanomatous skin lesion or carcinoma in situ of the cervix.
* Patient must not have Acquired Immune Deficiency Syndrome (AIDS) or HIV positive based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS or HIV from this protocol is necessary because anti-retrovirals may alter patient metabolism.
* Patient may not have any active Gastrointestinal/Malabsorption disorder at the discretion of the Principal Investigator which may include:
* Chronic Pancreatitis
* Chronic Diarrhea or Vomiting
* Active Eating Disorder
* No history of or current active drug/alcohol dependence.
* No patients with decisional impairment.

Exclusion Criteria:

* Patient is male.
* Age <18 years
* Clinical stage IV cancer
* Inflammatory breast cancer (T4d)
* Women of childbearing potential with a positive serum beta hCG.
* Decision impaired patients.
* BMI < 21
* Weight < 120lbs
* Weight loss ≥10% in the last 3 mos
* Prior invasive non-breast malignancy (except non-melanomatous skin cancer, carcinoma in situ of the cervix) unless disease free for a minimum of 1 year prior to registration
* Non-epithelial breast malignancies such as sarcoma or lymphoma
* Active Gastrointestinal/Malabsorption disorder at the discretion of the Principal -Investigator which may include:

  * Chronic Diarrhea or Vomiting
  * Active Eating Disorder
  * Active drug/alcohol dependence or abuse history.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response assessed in tissue | At time of definitive breast surgery
  The portion of patients who adhere to the diet restriction will be computed along with a 95% exact confidence. An exact binomial test (with a onesided alpha of 0.05) will also be used to test whether adherence is greater than 60%.
Incidence of adverse events evaluated by CTCAE version 4.0 | Up to 24 months

SECONDARY OUTCOMES:
Number of study participants who receive the dietary intervention to the historical controls | Up to 24 months
  Will be compared to historical controls. Will be based on logistic regression, which will control for patient characteristics and clinical factors. The study has 81% power to detect an odds ratio of about 0.25 using a 2-sided alpha of 0.05
Weight changes | Up to 24 months
  Will be assessed by modeling body mass index as a function of time via mixed-effects regression.
Change in insulin | Up to 24 months
  Will be assessed as a function of time via mixed-effects regression.
Change in serum | Up to 24 months
  Will be assessed as a function of time via mixed-effects regression.
Distant metastases | Up to 24 months
  Will be analyzed via the Kaplan-Meier method and the logrank test.
Progression-free survival | Up to 24 months
  Kaplan-Meier curves will be generated and a log-rank value will be calculated.
Overall survival | Up to 24 months
  Will be analyzed with the Kaplan-Meier method and Cox proportional hazards regression.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Simone, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson Univeristy, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/